CLINICAL TRIAL: NCT06346847
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Clinical Study to Assess Effects of Postbiotic vs. Placebo in Participants With Moderate to Severe Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: Study to Assess Effects of Postbiotic vs Placebo in Participants With Diarrhea-predominant IBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A-Mansia Biotech S.A. (Industry)
Collaborators: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAC/231001/AKM/IBS
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Diarrhea-Predominant Irritable Bowel Syndrome
Keywords: IBS

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Postbiotic (Experimental): 1 capsule a day, 15 minutes before breakfast with a glass of water for 12 weeks
  Interventions: Dietary Supplement: Postbiotic
- Placebo (Placebo Comparator): 1 capsule a day, 15 minutes before breakfast with a glass of water for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Postbiotic — 1 capsule a day, 15 minutes before breakfast with a glass of water for 12 weeks
  Arms: Postbiotic
Dietary Supplement: Placebo — 1 capsule a day, 15 minutes before breakfast with a glass of water for 12 weeks
  Arms: Placebo

SUMMARY:
The present study is a randomized, double-blind, placebo-controlled, parallel group clinical study that assesses the effect of postbioc on the complaints of subjects with moderate to severe diarrhoea-predominant irritable bowel syndrome (IBS-D). The trial is also evaluating the potential of postbiotic on anxiety, low mood and stress of the participants, as well as its safety and tolerability.

The intervention duration for all the study participants is 12 weeks (intervention phase). Subsequently, the participants will be invited to return to site for an end of study assessment after 21 days of no intervention (post-intervention phase).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18 to 55 years old.
2. Individuals diagnosed for IBS within the last two years, and meets Rome-IV criteria for IBS: recurrent abdominal pain on average ≥1 day/week in ≥3 months prior to study (with symptom onset ≥6 months prior to study), associated with ≥2 of the following criteria:

   1. Related to defecation
   2. Associated with a change in frequency of stool
   3. Associated with a change in form (appearance) of stool.
3. Has IBS-D, i.e., more than ¼ (25%) of bowel movements with Bristol stool types 6 or 7 and less than ¼ (25%) of bowel movements with Bristol stool types 1 or 2); in other words, put practically and as per FDA: at least 2 days per week with at least one stool that has a consistency of Type 6 or Type 7 BSS.
4. Has an IBS-SSS of at least 175 points at screening.
5. Individuals either with abdominal pain or discomfort (≥ 6 to ≤ 10 on an 11-point scale).
6. Has had no prior line of conventional intervention for IBS or dietary change in the last 4 weeks before screening (e.g., low FODMAP, soluble fibers, antispasmodics, laxatives, obstipants, serotonin agonist/antagonist) i.e., recently diagnosed individuals
7. Individuals' agreement to comply with study procedures, in particular:

   1. to take IP as recommended,
   2. to avoid the use of other products which may influence the gastrointestinal (GI) complaints, mental symptoms or commensal flora during the study as defined in Section 6.8 Prior and Concomitant Therapy,
   3. to keep the habitual dietary habits, level of physical activity as well as the level of caffeine or nicotine (if any),
   4. to complete the individual's diary and study questionnaires.
8. Women of childbearing potential:

   1. commitment to use contraception methods,
   2. Negative pregnancy testing (beta human chorionic gonadotropin test in urine).
9. Readiness not to participate in another clinical study during this study.
10. Participation is based upon written informed consent by the individual following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product.
2. Smokers
3. Lactose or fructose intolerance.
4. Individuals with uncontrolled hypertension as assessed by systolic blood pressure ≥ to 160 mmHg and diastolic blood pressure ≥ to 100mmHg.
5. History of diverticulitis, intestinal obstruction, stricture, toxic megacolon, GI (gastro-intestinal) perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (e.g., aorto-iliac disease) or recent unexplained GI bleeding within 3 months prior to screening.
6. History of malignancy within 3 years before screening (except squamous and basal cell carcinomas and cervical carcinoma in situ).
7. History and/or presence of acute or chronic significant GI disease or digestion/absorption disorders (e.g., inflammatory bowel disease, coeliac disease, Clostridium difficile colitis, pancreatitis, disorders in digestive tract motility, gluten enteropathy, etc.)
8. Major gastric, hepatic, biliary, pancreas or intestinal surgery within the last 6 months prior to screening or planned during the study (appendectomy, hemorrhoidectomy, or polypectomy allowed as long as occurred > 3 months prior to study screening; uncomplicated laparoscopic or open cholecystectomy is allowed if no history of post-operative biliary tract pain and surgery occurred > 3 months prior to screening).
9. Clinically significant findings in colonoscopy within the 3 years prior to study.
10. Family history among first degree relatives of colorectal cancer or inflammatory bowel disease.
11. Individuals diagnosed with psychiatric disease (e.g., bipolar disorder, Schizophrenia) with or without medication in the last three years.
12. Individuals currently on medication for anxiety and/or depression
13. Individual has a history and/or presence of other clinically significant condition/disorder, which per investigator's judgement could interfere with the results of the study or the safety of the participants, e.g.:

    1. thyroid gland disorder
    2. hypertension
    3. diabetes mellitus
    4. eating disorder
    5. immunodeficiency
    6. relevant gynecological or urological disorder
    7. any other relevant serious organ or systemic diseases ( e.g., cardiovascular, respiratory, liver, renal, neurological disease, etc.)
14. Regular medication and/or supplementation within the last month prior to and planned during the study:

    1. antibiotics, probiotics, prebiotics within 4 weeks before enrollment for screening.
    2. medication for IBS complaints, e.g., bile acid binders (cholestyramine), rifaximin, alosetron, lubiprostone, eluxadoline and linaclotide
    3. which could influence gastrointestinal functions (e.g., laxatives, opioids, systemic corticosteroids, anti-cholinergics, anti-diarrheals, proton pump inhibitors, H2-blockers, etc.) as per investigator judgement. Exception: ad hoc use of Macrolits.
15. Regular use of psychopharmaca (e.g., hypnotics / sedative drugs, anxiolytics, antidepressants, neuroleptics, anticonvulsants) within 3 months prior to study or adaptogens (e.g., ginseng, Ashwagandha, satavari, St. John's Wort) within 6 weeks prior to and during the study.
16. Introductions of a specific diet (e.g., low carb, vegan, high fibre, low FODMAP) within last 3 months prior to and during the study.
17. Women of child-bearing potential: pregnancy or nursing.
18. History of or current abuse of drugs, alcohol, tobacco/nicotine or medica tion.
19. Participation in another study during the last 30 days prior to and during the study.
20. Any other reason for exclusion as per investigator's judgment, e.g., insufficient compliance with study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of Investigational Product relative to placebo on percentage responders in terms of improvement of the IBS-Symptom Severity Scores (SSS) in participants with moderate to severe diarrhea-predominant irritable bowel syndrome. | Baseline (Day 0), and Week 12 (Day 84)
  A responder is defined as a participant who has a decrease in IBS-SSS of at least 50 points (minimal clinically important difference or MCID)

SECONDARY OUTCOMES:
To assess the impact of the Investigational Product in comparison to placebo on the percentage of participants who are responders in terms of improvement of the IBS-SSS from baseline at week 8 | Baseline (Day 0) and Week 8 (Day 56)
  A responder is defined as a participant who has a decrease in IBS-SSS of at least 50 points (minimal clinically important difference or MCID)
To assess the impact of the Investigational Product in comparison to placebo on mean change in Generalized Anxiety Disorder (GAD)-7 score | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  The GAD-7 scores are calculated by assigning scores of 0, 1, 2, and 3 to the response categories. GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety and 15-21: severe anxiety. The change from baseline in GAD#7 scores will be assessed.
To assess the impact of the Investigational Product in comparison to placebo on the percentage of participants who are responders in terms of improvement of the GAD-7 from baseline at week 12. | Baseline (Day 0) and Week 12 (Day 84)
  The GAD-7 scores are calculated by assigning scores of 0, 1, 2, and 3 to the response categories. GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety; 5-9: mild anxiety; 10-14: moderate anxiety and 15-21: severe anxiety. The change from baseline in GAD#7 scores will be assessed. A decrease in GAD-7 of at least 4 points compared to baseline is considered clinically meaningful improvement.
To assess the impact of the Investigational Product in comparison to placebo on mean change in Patient Health Questionnaire (PHQ)-9 score | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  The PHQ-9 is the 9-item depression module. As a severity measure, the PHQ-9 score can range from 0 to 27. The score will be interpreted as follows: 0-4: None - Minimal 5-9: Mild 10-14: Moderate 15-19: Moderately severe 20-27: Severe
To assess the impact of the Investigational Product in comparison to placebo on the percentage of participants who are responders in terms of improvement of the PHQ-9 from baseline at week 12. | Baseline (Day 0) and Week 12 (Day 84)
  The PHQ-9 is the 9-item depression module. As a severity measure, the PHQ-9 score can range from 0 to 27. The score will be interpreted as follows: 0-4: None - Minimal 5-9: Mild 10-14: Moderate 15-19: Moderately severe 20-27: Severe. . A decrease in PHQ-9 of at least 2 points compared to baseline.
To assess the impact of the Investigational Product in comparison to placebo on mean change in Perceived Stress Scale (PSS) | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  The questions in this scale ask about feelings and thoughts of an individual during the last month.Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
To assess the impact of the Investigational Product in comparison to placebo on mean change in Bristol Stool Form Score (BSFS) | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  BSFS is expressed as decrease in the % of abnormal stool consistencies (and thus increase in the % with normal consistency).
To assess the impact of the Investigational Product in comparison to placebo on occurrence of normal BSFS score at the end of the study | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  BSFS is expressed as decrease in the % of abnormal stool consistencies (and thus increase in the % with normal consistency).
To assess the impact of the Investigational Product in comparison to placebo on the quality of life as assessed by the mean change in IBS-QOL scores | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  It measures 8 disease-relevant domains: dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual and relationship issues. It is a 34#item questionnaire with each item rated on a 5# point scale (34-170), with increasing scores indicating the deteriorating quality of life.
To assess the impact of the Investigational Product in comparison to placebo on mean change in IBS-SSS value | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  A responder is defined as a participant who has a decrease in IBS-SSS of at least 50 points (minimal clinically important difference or MCID)
To assess the impact of the Investigational Product in comparison to placebo on compliance with the intake of the investigational product | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  A diary will be provided to the participant for ensuring compliance. The participant will be asked to fill IP missed or lost details in the diary.
To assess the impact of the Investigational Product in comparison to placebo on Safety and tolerance | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  Adverse events, Vital signs (Pulse Rate, Blood Pressure), Liver Function test, Renal Function Test, Complete Blood Count
To assess the impact of the Investigational Product in comparison to placebo on the impact of IBS on their quality of life using the IBS-Quality of Life (IBS-QoL) instrument. | Baseline (Day 0), Week 4 (Day 28), Week 8 (Day 56), Week 12 (Day 84), Week 15 (Day 105)
  It measures 8 disease-relevant domains: dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual and relationship issues. It is a 34#item questionnaire with each item rated on a 5# point scale (34-170), with increasing scores indicating the deteriorating quality of life. A decrease of 10 points or more is considered a clinically meaningful improvement.

CONTACTS AND LOCATIONS:
Locations (23):
- India (23):
  - HCG Hospital, Ahmedabad, Gujarat
  - Anand Multispeciality Hospital, Vadodara, Gujarat
  - Stress Test Clinic, Mumbai, Maharashtra
  - Criticare Asia Multispeciality Hospital & Research Centre, Mumbai, Maharashtra
  - Surya Multispeciality Hospital, Nashik, Maharashtra
  - Astha Clinic, Nashik, Maharashtra
  - Apollo Hospital, Navi Mumbai, Maharashtra
  - Swara Hospital, Pālghar, Maharashtra
  - Gastrohub Hospital, Pune, Maharashtra
  - Umarji Mother and Child Care Hospital, Pune, Maharashtra
  - Lifeline Multispeciality Hospital, Pune, Maharashtra
  - Asian Institute of Medical sciences, Thane, Maharashtra
  - Maharaja Agrasen Superspeciality Hospital, Jaipur, Rajasthan
  - Samvedna Hospital, Varanasi, Uttar Pradesh
  - GCS Medical College, Hospital & Research Centre, Gujarat
  - Nand Hospital, Gujarat
  - Maharaja Agrasen Superspeciality Hospital, Jaipur
  - Birch Multispeciality Hospital, Maharashtra
  - Lifeline multispeciality hospital, Maharashtra
  - Astha Clinic, Nashik
  - Mata Roop Rani Maggo Hospital & IVF Center, New Delhi
  - Ford Hospital, Uttar Pradesh
  - Human care hospital, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No